CLINICAL TRIAL: NCT06355830
Title: Intermediate Age-related Macular Degeneration - Multimodal Analysis and Longitudinal Study
Acronym: Imaging4iAMD
Status: Recruiting | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: iNOVA4Health, NOVA Medical School|Faculdade de Ciências Médicas, NMS|FCM, UNL (Unknown); Centro Hospitalar de Lisboa Central EPE, Lisboa, Portugal (Unknown); Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Sponsor
Other Study IDs: RETimaging4iAMD
Record Dates: First submitted 2023-03-07; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Intermediate AMD; Progression Biomarkers; Late AMD; SD-OCT
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intermediate AMD: Subjects over 55 years old with drusen secondary to intermediate AMD
  Interventions: Diagnostic Test: Orthoptic assessment (Outcome measure)

INTERVENTIONS:
Diagnostic Test: Orthoptic assessment (Outcome measure) — The protocol image assessment is non-invasive and includes retinal imaging by Color Fundus photography (CFP), Spectral Domain Optical Coherence Tomography (SD-OCT), OCT-Angiography (OCT-A) using Spectralis OCT, with OCT Angiography Module (Heidelberg Eng. GmbH, Germany).

SUMMARY:
Study: observational prospective clinical study. Study population: Subjects over 55 years old with drusen secondary to intermediate AMD.

Recruitment: at the Medical Retinal Consultation from the Ophthalmology Department of CHULC.

Primary outcome: Identifying imaging predictors of iAMD progression.

DETAILED DESCRIPTION:
Individuals will be included consecutively and undergo retinal imaging including Color Fundus photography (CFP), Spectral Domain Optical Coherence Tomography (SD-OCT), OCT-Angiography (OCT-A) using Spectralis OCT, with OCT Angiography Module (Heidelberg Eng. GmbH, Germany), in order to characterize:

A. FUNDUS AUTOFLUORESCENCE

1. Analyse the correlation between drusen morphology and autofluorescent findings
2. Analyse the correlation between outer retinal layers morphology and autofluorescent findings
3. Assess anatomic biomarkers of disease progression

B. VASCULAR FINDINGS

1. Test if choriocapillaris perfusion is disturbed in Intermediate AMD patients;
2. Test if retinal capillary plexus perfusion is disturbed in Intermediate AMD patients:

   2.1. Analyze superficial retinal capillary plexus (SCP), 2.2. Analyze deep retinal capillary plexus (DCP);
3. Assess if choroidal and retinal vascular changes are related to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* To verify the existence of drusen secondary to intermediate AMD; Soft, cuticular and reticular pseudo-drusen will be considered.
* Accept and sign the consent.

Exclusion Criteria:

* Patients are excluded if it is not possible to obtain good quality CFP, SD-OCT, OCT-A images, if refractive error is ≥±6D or if there is any evidence of accumulation of extracellular fluid, haemorrhage, exudates or fibrosis.
* Additional exclusion criteria included any history of retinal surgery including laser treatment, signs of diabetic retinopathy, history of retinal vascular occlusion, history of anti-VEGF treatment in the study eye or any signs or history of hereditary retinal or macular dystrophy.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 55 years old with drusen secondary to intermediate AMD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in incomplete retinal pigment epithelial and outer retinal atrophy (iRORA) from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  iRORA is measured in μm
Change in Drusen morphology from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Drusen classified as Serous, Reticular or both
Change in Subfoveal drusen area from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Subfoveal drusen area is measured in μm2, based on SD-OCT Spectralis Heidelberg
Change in other drusen area from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Other drusen area is measured in μm2, based on SD-OCT Spectralis Heidelberg
Change in Drusen reflectivity from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Drusen reflectivity classified as a) Low, b) Intermediate, c) High
Change in other Drusen homogeneity from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Drusen homogeneity classified in a) Low b) Intermediate or c) High
Change in ellipsoid zone disruption from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  ellipsoid zone disruption changes classified in a) Yes or b) No
Change in Drusen homogeneity from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Drusen homogeneity classified as a) Homogeneous or b) Heterogeneous
Change in hyperreflective foci from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Hyperreflective foci changes classified in a) Yes or b) No
Change in hyperreflective foci location (within 500-μm disc area) from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  hyperreflective foci location (within 500-μm disc area) changes classified as a) Yes or b) No
Change in hyperreflective foci association to drusen from baseline | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  hyperreflective foci association to drusen from baseline classified as a) Yes or b) No
Progression to Moderate Vision Loss | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Progression defined as a decrease in ETDRS BCVA score of 15 or more letters.
Geographic Atrophy (GA) Growth Rate | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  The annual growth rate of GA or nascent GA area measured in square root transform of the area measured in mm2 (final values in mm), based on SD-OCT Spectralis Heidelberg

SECONDARY OUTCOMES:
Progression to Advanced AMD according to international classification/grading system | Months 0 (baseline), 6, 12, 18, 24, 30, 36, 42 and 48
  Progression defined as the development of geographic atrophy or choroidal neovascularization detected by OCT imaging using autofluorescence, infrared, and/or angiography modules.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Flores, MD, Principal Investigator — Centro Hospitalar Universitário de Lisboa Central, iNOVA4Health Nova Medical School, Universidade Nova de Lisboa; Sandra Tenreiro, PhD, Study Chair — iNOVA4Health Nova Medical School, Universidade Nova de Lisboa
Locations (1):
- Ophthalmology Service, Centro Hospitalar de Lisboa Central EPE, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No